CLINICAL TRIAL: NCT06153420
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of CIN-103 in Adults With Irritable Bowel Syndrome With Predominant Diarrhea (IBS-D)
Brief Title: Study of the Research Medicine CIN-103 in Adults With Irritable Bowel Syndrome With Predominant Diarrhea (IBS-D).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy compared to placebo.
Sponsor: CinPhloro Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIN-103-121
Record Dates: First submitted 2023-11-09; First posted 2023-12-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; IBS-D; IBS; IBS with diarrhea; Abdominal pain with diarrhea; IBS with loose stool
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CIN-103 BID Dose 1 (Experimental): CIN-103 Dose 1, administered as 2 x CIN-103 capsules and 2 x matching placebo per dose. Two doses per day.
  Interventions: Drug: CIN-103
- CIN-103 BID Dose 2 (Experimental): CIN-103 Dose 2, administered as 4 x CIN-103 capsules per dose. Two doses per day.
  Interventions: Drug: CIN-103
- Placebo for CIN-103 BID (Placebo Comparator): Placebo for CIN-103, administered as 4 x matching placebo capsules per dose. Two doses per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-103 — CIN-103 BID
  Arms: CIN-103 BID Dose 1; CIN-103 BID Dose 2
Drug: Placebo — Placebo for CIN-103 BID
  Arms: Placebo for CIN-103 BID

SUMMARY:
The goal of this clinical trial is to evaluate if the study drug, CIN-103, can help reduce the symptoms associated with irritable bowel syndrome with predominant diarrhea (IBS-D) in adult patients. The main questions it aims to answer are:

* To evaluate the efficacy of CIN-103 on symptoms of IBS-D when given to patients with IBS-D compared to a placebo.
* To evaluate the safety and tolerability of CIN-103 when given to patients with IBS-D compared to a placebo

Participants will attend the following visits:

* Screening Period (1 Visit)
* Baseline Period (1 Visit)

  * Will complete daily diary and other Patient Reported Outcomes (PROs) as described in the protocol to assess eligibility for continued participation.
* 12-Week Treatment Period (5 Visits)

  * Study drug taken twice daily by mouth.
  * Will complete daily diaries and other PROs as described in the protocol.
* Follow- Up Period (1 Visit)

Researchers will compare CIN-103 Dose 1, CIN-103 Dose 2, and placebo, to evaluate the clinical response to multiple dose strengths of CIN-103 relative to placebo on abdominal pain and stool consistency along with safety and tolerability.

ELIGIBILITY:
* Inclusion Criteria:

  1. Are adult male and female subjects ≥ 18 years of age;
  2. Have a body mass index between 18 and 45 kg/m2, inclusive at Screening;
  3. Meet Rome IV Criteria for IBS-D by subject self-report of recurrent abdominal pain that is associated with ≥ 2 of the following over the last ≥ 6 months, with frequency of at least 1 day per week over the last 3 months (on average) before enrollment:

     1. Related to defecation;
     2. Associated with a change in frequency of stool; and/or
     3. Associated with a change in form (appearance of stool).
  4. Based on Investigator interview of subject's symptoms over the last 3 months, have ≥ 25% of bowel movements (BMs) with Bristol Stool Scale (BSS) Type 6 or 7 (loose or watery stools) and < 25% of BMs with BSS Type 1 or 2 (lumpy or hard stools) per the Rome IV Criteria for IBS-D;
  5. In the opinion of the Investigator, are on a stable diet for ≥ 4 weeks prior to Screening and are not planning to change lifestyle, exercise, and/or diet that may impact symptoms of IBS-D during study participation;
  6. Have a fecal calprotectin ≤ 100 mcg/g at the Screening Visit or Visit 2; Note: A single normal test result is adequate for study eligibility. If subjects are rescreened within 12 months, there is no need for repeat fecal calprotectin sample collection and testing. However, subjects who fail screening due to a fecal calprotectin level > 100 mcg/g are not eligible for re-screening. Note: Repeat Fecal calprotectin may be considered with prior Sponsor approval.
  7. Have a serum tTG-IgA (tissue transglutaminase immunoglobulin A) ≤ 4.99 FLU (fluorescent light units) at the Screening Visit;
  8. Have undergone a colonoscopy examination within the designated time interval prior to randomization, if they meet any of the following criteria. Note: A negative Cologuard® test result is an acceptable alternative to colonoscopy for subjects ≥ 45 years and at average risk for colon cancer.

     1. Average risk, based on US Preventive Services Task Force Recommendation Statement for screening of colorectal cancer, with age ≥ 45 years (colonoscopy within 10 years or negative test results on Cologuard within 3 years);
     2. Personal history of completely removed adenomatous colorectal polyps (colonoscopy within 5 years for polyps > 1 cm, within 10 years for polyps < 1 cm);
     3. History of colorectal cancer or adenomatous polyps in a first-degree relative before age 60 (colonoscopy within 5 years); or
     4. History of colorectal cancer or adenomatous polyps in ≥ 2 first-degree relatives at any age, or family history of hereditary colorectal cancer or polyposis (colonoscopy within 5 years).
* Exclusion Criteria:

  1. Have a diagnosis or suspected diagnosis of non-diarrhea predominant IBS (eg, IBS with a subtype of constipation, IBS with mixed or alternating bowel habits, un-subtyped IBS) or functional constipation by the Rome IV Criteria;
  2. Non-infectious chronic lower gastrointestinal conditions including a history of or current inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis, indeterminate colitis), recurrent diverticulitis, microscopic colitis, lymphocytic colitis, celiac disease, non-celiac gluten sensitivity and non-compliant on a gluten-free diet, untreated lactose intolerance, carcinoid syndrome, Lynch syndrome, or familial polyposis, intestinal obstruction, stricture, toxic megacolon, solitary rectal ulcer syndrome, GI perforation, intra-abdominal or pelvic adhesions, ischemic colitis, radiation proctitis, chronic enteritis, non-infectious colitis, or impaired intestinal circulation (eg, aortoiliac disease);

     Note: Lactose intolerance and non-celiac gluten sensitivity will not exclude a subject from participation if the Investigator documents that the subject is compliant on a special diet (lactose-free diet or gluten-free diet, respectively) and/or for lactose intolerance is successfully treated with commercial lactase supplement(s).
  3. Infectious lower gastrointestinal conditions requiring antibiotics or microbiome therapy; any microbiologically documented acute lower gastrointestinal colitis or enteritis requiring antibiotic treatment including successfully treated Clostridioides difficile colitis within 3 months prior to Screening, or a history of recurrent C. difficile colitis at any time in the past;
  4. Have a known family history of inflammatory bowel disease in at least 1 first-degree relative;
  5. Have a known history of a pelvic floor disorder associated with constipation (unless successful treatment has been documented by a normal balloon expulsion test or anorectal manometry), refractory constipation not responsive to standard medical therapy, fecal impaction that required hospitalization, cathartic colon, and/or active proctological condition;
  6. Have a history of or current non-IBS chronic condition(s) with ongoing symptoms associated with abdominal pain or GI discomfort (eg, gastroparesis, functional dyspepsia, uncontrolled gastroesophageal reflux disease, polycystic kidney disease, ovarian cysts, urological pain, or endometriosis);
  7. Have a history of or current clinically significant arrhythmias as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, and Torsades de pointes. Subjects with any abnormal electrocardiogram (ECG) not considered clinically significant by the Investigator are not excluded;
  8. Have current or a history of diverticulitis, heme positive stool, or unexplained GI bleeding within 3 months prior to Screening.

     Note: Surgically repaired diverticulitis > 3 months prior to Screening is permitted.
  9. Have a history of surgical resection of the stomach, small, or large intestine;
  10. Have had any major abdominal surgery within the 3 months prior to Screening;

      Note: Permitted procedures are uncomplicated appendectomy, cholecystectomy, and resection of benign polyps within the 3 months prior to Screening. Subjects who had an appendectomy that was associated with any related complications or sequelae are eligible if the procedure was performed at least 6 months prior to Screening.
  11. Are currently undergoing or planning to initiate treatment with weight loss medication during study participation or prior weight loss surgery (eg, gastric bypass surgery, gastric banding);
  12. Have a planned invasive elective surgery during the period of anticipated study participation from the time of informed consent through the last study visit;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of meeting Study Composite Responder status for an adult subject with IBS-D. | 12 weeks of Double Blind Treatment Period
  A subject is defined as a Study Composite Responder if he or she meets the Daily Composite Responder criteria for at least 50% of days with diary entry during the 12-week Double-Blind Treatment Period. A subject is defined as a Daily Composite Responder if he or she meets both the pain intensity and stool consistency criteria as follows:
  * Improvement in the mean daily worst abdominal pain (WAP) score by ≥ 30% compared to the mean daily WAP score from the Baseline Period (the average of the daily measurements over the 14 days prior to randomization); AND
  * Improvement in stool consistency based on the Bristol Stool Scale (BSS) score < 5 or the absence of a bowel movement (BM) over the past 24 hours.
  Note: If a subject did not have a BM, an improvement of at least 30% in the WAP score is sufficient for a response on that day.
  The proportion of subjects with a primary outcome within each dose of CIN-103 will be compared to the proportion of subjects in the placebo arm.

SECONDARY OUTCOMES:
The occurrence of meeting Weekly Composite Responder status | 12-week of Double-Blind Treatment Period
The occurrence of meeting Weekly Composite Responder status over 4-weekly intervals (1 to 4, 5 to 8, and 9 to 12 weeks). | 12 weeks of Double Blind Treatment Period
  A subject is defined as a Weekly Composite Responder if he or she meets both abdominal pain and stool consistency criteria as follows: An Abdominal Pain Intensity Weekly Responder is defined as a subject who experiences a decrease in the weekly average of WAP in the past 24 hours score of at least 30% compared with Baseline; AND A Stool Consistency Weekly Responder is defined as a subject who experiences a 50% or greater reduction in the number of days per week with at least 1 stool that has a consistency of Type 6 or 7 compared with Baseline.
The change in a composite of the daily mean and weekly mean of daily WAP score and stool consistency score as compared to Baseline | 12-week of Double-Blind Treatment Period
  The subject-reported WAP in the past 24 hours will be recorded on an 11-point (ie, 0 to 10) numeric rating scale, where 0 corresponds to no pain and 10 corresponds to worst imaginable pain. The stool consistency will be measured using the Bristol Stool Score, based on a 1 to 7 scale where 1 corresponds to a hard stool and 7 corresponds to watery diarrhea.
The change in daily mean and weekly mean number of BMs per day compared to Baseline | 12-week of Double-Blind Treatment Period
The occurrence of meeting Stool Consistency Responder status | 12-week of Double-Blind Treatment Period
  A participant is considered a Stool Consistency Responder if there is an improvement in stool consistency based on the BSS score < 5 or the absence of a bowel movement over the past 24 hours.
The change in the daily mean and weekly mean of stool consistency measured with the Bristol Stool Scale (BSS) as compared to Baseline | 12-week of Double-Blind Treatment Period
  The subject-reported BSS consistency score is based on a 1 to 7 scale where 1 corresponds to a hard stool and 7 corresponds to watery diarrhea.
The occurrence of meeting Pain Responder status | 12-week of Double-Blind Treatment Period
  A participant is considered a Pain Responder if there is an improvement in the mean daily WAP score by ≥ 30% compared to the mean daily WAP score from the Baseline Period (the average of the daily measurements over the 14 days prior to randomization).
The change in the daily mean and weekly mean of daily WAP as compared to Baseline | 12-week of Double-Blind Treatment Period
The change in the daily mean and weekly mean of daily abdominal bloating score as compared to Baseline. | 12-week of Double-Blind Treatment Period
  The subject-reported abdominal bloating in the past 24 hours will be recorded on an 11-point (ie, 0 to 10) numeric rating scale, where 0 corresponds to no bloating and 10 corresponds to worst imaginable bloating.
The change in the daily mean and weekly mean of daily urgency score compared to Baseline. | 12-week of Double-Blind Treatment Period
  Daily urgency score is measured on a numeric rating scale from 0 (no urgency) to 10 (worst possible urgency).
The change in daily mean and weekly mean number of fecal incontinence episodes compared to Baseline | 12-week of Double-Blind Treatment Period
  Subjects will receive daily automatic reminders on eDiary to record the number of fecal incontinence episodes over the past 24 hours.
Incidence of clinically significant changes, in the Investigator's opinion, in vital signs, physical examinations, ECGs, and clinical laboratory evaluations. | Through study completion, up to 19 weeks.
  Including standard safety chemistry panel, hematology, coagulation, lipids, and urinalysis.
Occurrence of Treatment-Emergent Adverse Events (TEAEs). | Through study completion, up to 19 weeks.
Occurrence of treatment-emergent serious adverse events. | Through study completion, up to 19 weeks.
Occurrence of TEAEs leading to premature discontinuation of the study drug. | Through study completion, up to 19 weeks.
Occurrence of treatment-emergent clinically significant laboratory abnormalities. | Through study completion, up to 19 weeks.
Percentage of post-randomization days with symptom of urgency present ("Yes") | 12-week of Double-Blind Treatment Period
  The severity of bowel urgency will be captured on a numeric rating scale from 0 (no urgency) to 10 (worst possible urgency). Using this scale, bowel urgency will also be captured as not present "No" (score 0) or present "Yes" (score 1 to 10).

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Digestive Health Specialists - Dothan, Dothan, Alabama
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - GI Alliance - Sun City, Sun City, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Paragon Rx Clinical, Inc. - Garden Grove, Garden Grove, California
  - Gastro Care Institute- lancaster, Lancaster, California
  - Medical Associates Research Group, San Diego, California
  - American Family Research Group, Cape Coral, Florida
  - USA and International Research Inc., Doral, Florida
  - International Research Associates LLC, Miami, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Velocity Clinical Research,, Savannah, Savannah, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - DelRicht Research, Mandeville, Louisiana
  - Tandem Clinical Research GI LLC, Marrero, Louisiana
  - Tandem Clinical Research GI LLC, Metairie, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Delta Research Partners, LLC, West Monroe, Louisiana
  - DelRicht Research of Bethesda Clinical Trials, Rockville, Maryland
  - St. Charles Clinical Research, Weldon Spring, Missouri
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Advanced Research Institute - Reno, Reno, Nevada
  - Allied Digestive Health Clinical Research Organization, Somers Point, New Jersey
  - Allied Digestive Health-Jersey Shore Gastroenterology - Point Commons, Somers Point, New Jersey
  - Albuquerque Clinical Trials, Inc, Albuquerque, New Mexico
  - Westchester Putnam Gastro, Carmel Hamlet, New York
  - IMA Clinical Research PC and Affiliates- New York, NY, New York, New York
  - NY Scientific, New York, New York
  - Atrium Health - Center for Gastroenterology and Hepatology MMP, Charlotte, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - IMA Clinical Research, Mount Airy, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Remington Davis, Inc., Columbus, Ohio
  - Great Lakes Gastroenterology Research LLC, Mentor, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Options Health Research LLC, Tulsa, Oklahoma
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - DelRicht Research of Charleston Clinical Trials, Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Galen Medical Group - Downtown Gastroenterology Location, Chattanooga, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - The Clinical Trials Network LLC, Houston, Texas
  - Care and Cure Clinic, Houston, Texas
  - GLRI - McAllen Research, Pharr, Texas
  - Quality Research Inc, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - GI Alliance - Washington Gastroenterology, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No